CLINICAL TRIAL: NCT03217773
Title: Endoscopic Submucosal Dissection (ESD) Versus Transanal Minimally Invasive Surgery (TAMIS) for Early Rectal Neoplasms: a Prospective Randomized Controlled Trial
Brief Title: ESD Versus TAMIS for Early Rectal Neoplasms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Simon S. M. Ng, Professor of Surgery, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CREC Ref. No.: 2016.680-T
Record Dates: First submitted 2017-07-12; First posted 2017-07-14 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Rectal Neoplasms
MeSH Terms: conditions — Rectal Neoplasms | interventions — Transanal Endoscopic Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESD (Experimental): ESD is an endoscopic procedure that enables en bloc resection of large tumors in the gastrointestinal tract, irrespective of the size of the lesion. ESD uses an electrosurgical cutting device to purposely dissect the deeper layers of the submucosa to remove neoplastic mucosal lesions in a single piece.
  Interventions: Procedure: ESD
- TAMIS (Active Comparator): TAMIS is a minimally invasive means of removing large rectal neoplastic lesions not accessible by conventional transanal excision. It is performed using the GelPOINT path transanal access platform and laparoscopic instruments.
  Interventions: Procedure: TAMIS

INTERVENTIONS:
Procedure: ESD — Refer to arm description
  Arms: ESD
Procedure: TAMIS — Refer to arm description
  Arms: TAMIS

SUMMARY:
This is a prospective randomized controlled trial that aimed to compare the short-term clinical outcomes, functional outcomes, costs, and recurrence rates between endoscopic submucosal dissection (ESD) and transanal minimally invasive surgery (TAMIS) for early rectal neoplasms.

DETAILED DESCRIPTION:
Background: Transanal minimally invasive surgery (TAMIS) is an effective surgical alternative to transanal excision for treating early rectal neoplasms not amenable to en bloc resection by conventional colonoscopic techniques. Endoscopic submucosal dissection (ESD) is a revolutionary endoscopic procedure that enables en bloc resection of large rectal neoplasms with low morbidity. To date, no randomized controlled trial can be found in the literature comparing the two modalities.

Objectives: To compare the short-term clinical outcomes, functional outcomes, costs, and recurrence rates between ESD and TAMIS for early rectal neoplasms.

Design: Prospective randomized controlled trial.

Subjects: One hundred and fourteen consecutive patients diagnosed with early rectal neoplasms (>/=2 cm in size and without evidence of deep submucosal invasion) that are not amenable to en bloc resection by conventional colonoscopic techniques will be recruited.

Interventions: Patients will be randomly allocated to receive either ESD or TAMIS.

Outcome measures: Primary outcome: 30-day morbidity/mortality defined by the Clavien-Dindo classification. Secondary outcomes: hospital stay, functional outcomes and quality of life, overall costs, R0 resection rate, and recurrence rate.

Conclusions: Results of the present study can provide evidence-based clarification of the efficacy and safety of ESD in treating early rectal neoplasms. The Investigators hypothesize that ESD is associated with lower morbidity, shorter hospital stay, and similar R0 resection rate when compared with TAMIS. A faster recovery and earlier discharge after ESD may reduce financial burden to the hospital/healthcare system. The results of this proposed project may have a significant impact on the future treatment strategy for early rectal neoplasms.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with nonpedunculated early rectal neoplasms >/= 2 cm in size in the rectum (>/= 3 cm and </= 18 cm from the anal verge) that are deemed not feasible for en bloc resection with conventional polypectomy or EMR as judged by two experienced endoscopist
* Age of patients >18 years;
* American Society of Anesthesiologists (ASA) grading I-III
* Informed consent available

Exclusion Criteria:

* Presence of endoscopic signs of massive submucosal invasion (including excavated/depressed morphology, Kudo's pit pattern Type V, or Sano's capillary pattern Type IIIB)
* Evidence of deep invasion on endorectal ultrasonography
* Unfavorable histopathologic features on biopsy (mucinous cancer, poor differentiation, or gross submucosal invasion)
* Patients with other synchronous colorectal neoplasms in addition to the index neoplasm that are indicated for surgical resection
* Patients with recurrence from previous Endoscopic Mucosal Resection or ESD
* Patients with known metastatic disease
* Patients with non-correctable coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Short-term morbidity | Up to 1 month
  Short-term morbidity/mortality within 30 days after the procedure (including intraprocedural morbidity/mortality), defined by the Clavien-Dindo classification of surgical complications

SECONDARY OUTCOMES:
En bloc resection rate | Up to 1 month
  Resection with a single piece
R0 resection rate | Up to 1 month
  Complete resection of the neoplasm with clear lateral and deep margins at histology
Time to resume normal diet | Up to 1 month
Time to walk independently | Up to 1 month
Length of hospital stay | Up to 1 month
Anal continence | Up to 1 year
  Measured by the Wexner's score
Fecal incontinence quality of life (FIQL) | Up to 1 year
  Measured by the FIQL questionnaire
Quality of life measured by the Short Form-36 (SF-36) Health Survey questionnaire | Up to 1 year
  SF-36 Health Survey is a 36-item, patient-reported survey of patient health. It consists of eight scaled scores, which are the weighted sums of the questions in their section. The eight sections are: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Direct medical costs | Up to 1 year
Local recurrence | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Simon SM Ng, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No